CLINICAL TRIAL: NCT03377816
Title: The Role of Emotional Processing in Improving the Quality of Life of Breast Cancer Patients: a Mechanistic Study of Art Therapy in Reducing Depression, Fatigue and Pain.
Brief Title: The Role of Emotional Processing in Improving the Quality of Life of Breast Cancer Patients
Acronym: REPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: University of Arizona (Other); Monash University (Other); Rabin Medical Center (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Johanna Czamanski-Cohen, Principal Investigator, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UHaiArtBC; R01NR017186 (NIH)
Record Dates: First submitted 2017-12-10; First posted 2017-12-19 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer Female; Depressive Symptoms; Fatigue; Pain; Emotions; Inflammation
Keywords: Emotion Processing; Art Therapy; Breast Cancer; Cholinergic anti-inflammatory pathway
MeSH Terms: conditions — Depression; Fatigue; Pain; Inflammation; Breast Neoplasms | interventions — Art Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The control group is designed to be similar to the intervention, participants will be engaged in interacting with art materials. Research assistants will be blinded to group allocation when collecting data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy (Experimental): The AT intervention is an 8-week group intervention comprised of 8 1.5 hour weekly sessions conducted by an experienced Art Therapist who received special training in conducting the treatment protocol as designed.
  Interventions: Behavioral: Art Therapy
- Mandala group (Sham Comparator): The comparison group will color prefabricated shapes. The same art materials as in the intervention group will be on the table as will the same instrumental music.
  Interventions: Behavioral: Sham Art Therapy

INTERVENTIONS:
Behavioral: Art Therapy — In a group setting participants will be encouraged to engage in art making for increased emotional awareness, expression, and acceptance. The role of the art therapist is to encourage a non-judgmental and exploratory approach to artmaking in which the process is emphasized over product. The art therapist obtains these goals by creating an atmosphere that is calm and by remaining tuned in to the verbalizations and body language of participants. If needed she can provide individual attention that is geared toward neutralizing concerns regarding performance during the art making.
  Arms: Art Therapy
Behavioral: Sham Art Therapy — In a group setting participants will engage in Mandala coloring
  Arms: Mandala group

SUMMARY:
The purpose of this study is to examine two mechanistic changes: emotion processing (awareness, expression and acceptance) and cholinergic anti-inflammatory processes (HRV and cytokine expression) through which an Art Therapy (AT) intervention reduces depression, pain and fatigue.

DETAILED DESCRIPTION:
The study is a randomized controlled study with careful controls. Our study population is comprised of 240 BC patients in palliative and curative care (comprised of 50% Jewish and 50% Arab). This population will be randomized to receive a standard art therapy intervention or a comparison group. The AT intervention is an 8-week group intervention comprised of 8 1.5 hour weekly sessions conducted by an experienced Art Therapist The comparison group will engage in the coloring of prefabricated shapes (mandalas) and will receive Psychoeducation on topics related to coping with BC, identical to the topics of the AT group. This design will allow the study to test the mechanism of AT that is beyond the effects of time with a group, focus on a task and engagement with art materials.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18) females with initial or recurrent BC
* intervention can begin 3 months after finishing chemotherapy and radiotherapy (RT) and one month after surgery, up until 18 months after treatment completion.
* can complete assessments in Arabic or Hebrew
* provides informed consent.

Exclusion Criteria:

* male
* lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder or with a pre- cancer diagnosis of fibromyalgia or chronic fatigue syndrome
* active suicidal plan (will ensure immediate intervention);
* dementia/other disorder that would preclude informed consent or comprehension of assessments
* Individuals taking anticholinergic medications, and post myocardial infarction (6 months before recruitment) or with a pacemaker, which would render the metric of HRV invalid.
* Flare-up in systemic autoimmune disease (such as arthritis, lupus or multiple sclerosis), thyroid dysfunction that requires increases in medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czamanski-Cohen J, Wiley J, Weihs KL. Protocol for the REPAT study: role of emotional processing in art therapy for breast cancer palliative care patients. BMJ Open. 2020 Nov 19;10(11):e037521. doi: 10.1136/bmjopen-2020-037521. PMID 33444178
- [Background] Czamanski-Cohen J, Weihs KL. The role of emotion processing in art therapy (REPAT) intervention protocol. Front Psychol. 2023 Jun 29;14:1208901. doi: 10.3389/fpsyg.2023.1208901. eCollection 2023. PMID 37457095
- See also: Related Info — https://repat.haifa.ac.il/en/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Art Therapy | Mandala Group
Started | 157 | 161
Completed | 107 | 108
Not Completed | 50 | 53

BASELINE CHARACTERISTICS:
Population: 318 BC survivors over the age of 18 signed informed consent and were randomized to one of two groups, 289 completed baseline measurements.
Groups:
- Total: Total of all reporting groups
Arm/Group | Art Therapy | Mandala Group | Total
Number analyzed (Participants) | 146 | 143 | 289
Age, Customized [Count of Participants; unit: Participants]
  Age: 26-35 | 9 | 5 | 14
  Age: 36-45 | 31 | 23 | 54
  Age: 46-70 | 80 | 85 | 165
  Age: 70+ | 9 | 9 | 18
  Age: missing | 17 | 21 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 143 | 289
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 146 | 143 | 289
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 146 | 143 | 289

OUTCOME MEASURES:

1. Primary Outcome: Depression Depression
Description: The Center for Epidemiologic Studies-Depression (CES-D) 10-item scale. The possible range of scores is zero to 50, with the higher scores indicating the presence of more symptomatology.
Time Frame: Changes will be measured from baseline (T1), after the intervention (8-10 weeks after baseline T2) and 8 weeks after the intervention ends (T3)
Population: The posted data are raw, before multiple imputations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Art Therapy | Mandala Group
Number analyzed (Participants) | 122 | 118
score on a scale
  T1 | 10.82 (6.01) | 11.57 (6.46)
  T2: number analyzed (Participants) | 80 | 75
  T2 | 9.86 (6.203) | 11.23 (5.45)
  T3: number analyzed (Participants) | 65 | 69
  T3 | 11.05 (5.67) | 11.72 (5.59)

2. Primary Outcome: Fatigue
Description: Fatigue will be assessed using the Fatigue Symptom Inventory (FSI), a 14-item self-report measure designed to assess the severity of fatigue on an 11-point scale (0=not at all fatigued; 10=as fatigued as I could be) that assesses most, least, and average fatigue in the past week. A global score can be obtained summing items 1-13, resulting in a scale with a range between 0-130. Higher results represent higher levels of global fatigue.
Time Frame: as for outcome 1
Population: We utilized full maximum likelihood, and the numbers presented here are raw data in which if an individual missed one item from the scale, it was marked as missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Art Therapy | Mandala Group
Number analyzed (Participants) | 117 | 120
score on a scale
  T1 | 61.35 (28.77) | 63.08 (29.69)
  T2: number analyzed (Participants) | 75 | 72
  T2 | 53.28 (29.4) | 58.99 (24.79)
  T3: number analyzed (Participants) | 59 | 67
  T3 | 60.36 (29.4) | 63.21 (28.38)

3. Primary Outcome: Pain (Impact and Interference)
Description: The PROMIS Pain impact Scale measures how much pain impacted different aspects of life in the past 7 days. Scores range from 0-to-60, higher scores indicating higher levels of pain or its impact on functioning and the PROMIS Pain Interference Scale measures how much pain interfered with different aspects of life in the past 7 days. Scores range from 0-to-60, higher scores indicating higher levels of pain or interference with functioning. Our data indicates t-scores calculated so that 50 indicates the population (cancer patient) mean with a standard deviation of 10.
Time Frame: as for outcome 1
Population: The overall number of participants analyzed reflects the number of participants at T1. We used the maximum likelihood analyses, thus each row reflects the actual number of participants who had full data and the respective means and standard deviations.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Art Therapy | Mandala Group
Number analyzed (Participants) | 124 | 118
t-score
  Pain intensity T1 | 58.74 (12.5) | 57.4 (12.3)
  Pain intensity T2: number analyzed (Participants) | 80 | 75
  Pain intensity T2 | 55.9 (11.9) | 56.1 (11.8)
  Pain intensity T3: number analyzed (Participants) | 65 | 69
  Pain intensity T3 | 59.1 (11.6) | 58.0 (12.5)
  Pain interference T1: number analyzed (Participants) | 123 | 118
  Pain interference T1 | 59.0 (9.3) | 59.3 (9.4)
  Pain interference T2: number analyzed (Participants) | 80 | 74
  Pain interference T2 | 56.7 (9.43) | 57.1 (9.0)
  Pain interference T3: number analyzed (Participants) | 65 | 69
  Pain interference T3 | 59.0 (9.0) | 57.7 (9.3)

4. Secondary Outcome: Emotional Awareness
Description: The Levels of Emotional Awareness Scale is a written performance index of ability to express emotion in a differentiated and complex way. Subjects write about their anticipated feelings and those of another person in response to 10 short vignettes. Responses are scored on a 1 - 4 range and summed up to create a range of 0-50 according to the degree of specificity in the terms used and the range of emotions described, higher scores indicating higher levels of awareness.
Time Frame: as for outcome 1
Population: We used maximum likelihood for analyses. The numbers here reflect raw data, where if one question was not answered, the whole questionnaire is marked as missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Art Therapy | Mandala Group
Number analyzed (Participants) | 114 | 110
score on a scale
  T1 | 30.11 (5.28) | 30.59 (6.24)
  T2: number analyzed (Participants) | 77 | 68
  T2 | 30.87 (4.523) | 30.9 (5.49)
  T3: number analyzed (Participants) | 59 | 64
  T3 | 30.12 (5.21) | 28.77 (4.84)

5. Secondary Outcome: Emotional Expression
Description: This is a 36-item scale in which participants respond on a Likert scale from 1 (I don't do this at all) to 4 (I do this a lot) regarding how they coped with breast cancer experiences in the past four weeks. Two subscales are created from means of items: Approach Coping composite (24 items), and Avoidance composite (12 items) each with a range from 1-4 . Higher scores indicate more approach-oriented or avoidance-oriented coping. Participants rated items on a response scale of 1 (''I don't do this at all'') to 4 (''I do this a lot'').
Time Frame: Changes will be measured from baseline (T1), after the intervention (8-10 weeks after baseline (T2), and 8 weeks after the intervention ends (T3)
Population: We utilized maximum likelihood, and here are presented raw data, in which if a participant missed one question, the data was marked as missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Art Therapy | Mandala Group
Number analyzed (Participants) | 106 | 98
score on a scale
  Approach T1: number analyzed (Participants) | 106 | 93
  Approach T1 | 3.2596 (0.44) | 3.185 (0.54)
  Approach T2: number analyzed (Participants) | 64 | 64
  Approach T2 | 3.17 (0.52) | 3.169312169 (0.52)
  Approach T3: number analyzed (Participants) | 54 | 54
  Approach T3 | 3.078 (0.48) | 3.21 (0.52)
  Avoidance T1 | 1.99 (0.56) | 2.08 (0.59)
  Avoidance T2: number analyzed (Participants) | 68 | 69
  Avoidance T2 | 2.04 (0.78) | 2.18 (0.7)
  Avoidance T3: number analyzed (Participants) | 57 | 59
  Avoidance T3 | 2.21 (0.67) | 2.27 (0.74)

6. Secondary Outcome: Acceptance of Emotions
Description: The Acceptance of Emotions Scale assesses the extent to which subjects are accepting and nurturing toward their feelings, ranging 0-100, higher scores indicate higher acceptance of emotion.
Time Frame: as for outcome 1
Population: We conducted maximum likelihood analyses and the numbers here are raw scores, in which if a participant skipped one item the entire questionnaire was marked missing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Art Therapy | Mandala Group
Number analyzed (Participants) | 123 | 119
score on a scale
  T1 | 67.7756 [48.14273 to 87.40847] | 63.8561 [39.8156 to 87.8966]
  T2: number analyzed (Participants) | 79 | 75
  T2 | 66.12 [41.852 to 90.753] | 68.42 [45.811 to 90.696]
  T3: number analyzed (Participants) | 65 | 69
  T3 | 69.86 [51.84674999 to 88.72084908] | 71.29713424 [50.35255616 to 92.24171231]

7. Secondary Outcome: Inflammation
Description: We collected 10 ccs of blood in order to measure immune regulation (pro-inflammatory cytokines IL-6, IL-8, IL-1β, TNF-α), anti-inflammatory (IL-4, IL-10) and regulatory cytokines (TGF-β).
Time Frame: Changes will be measured from baseline (T1), after the intervention, 8-10 weeks after baseline T2) and 8 weeks after the intervention ends (T3).
Population: Number in each row reflect the number of results obtain for each cytokine at each time point. The overall number analyzed reflects the largest number of individuals that provided blood that was able to produce a quantification of at least one cytokine.
Measure: Mean (Standard Deviation); unit: pcg/ml
Arm/Group | Art Therapy | Mandala Group
Number analyzed (Participants) | 117 | 110
pcg/ml
  IL-8 T1: number analyzed (Participants) | 117 | 108
  IL-8 T1 | 15.78 (24.3) | 22.1597 (55.01)
  IL-8 T2: number analyzed (Participants) | 69 | 67
  IL-8 T2 | 11.02 (10.65) | 11.84 (11.9)
  IL-8 T3: number analyzed (Participants) | 51 | 54
  IL-8 T3 | 9.0135 (7.725) | 9.278 (9.38)
  il_1b_T1: number analyzed (Participants) | 117 | 105
  il_1b_T1 | 0.42 (1.15) | 0.55 (1.37)
  il_1b_T2: number analyzed (Participants) | 68 | 66
  il_1b_T2 | 0.18 (0.312) | 0.227 (0.5)
  il_1b_T3: number analyzed (Participants) | 50 | 52
  il_1b_T3 | 0.2632 (0.77) | 0.234 (0.68)
  il_4_T1: number analyzed (Participants) | 101 | 98
  il_4_T1 | 16.8 (31.6) | 24.33 (50.3)
  il_4_T2: number analyzed (Participants) | 66 | 59
  il_4_T2 | 10.1 (17.53) | 12.7 (23.09)
  il_4_T3: number analyzed (Participants) | 48 | 50
  il_4_T3 | 11.2 (35.7) | 14.58 (40.49)
  il_6_T1: number analyzed (Participants) | 117 | 105
  il_6_T1 | 1.4 (3.1) | 1.52 (3.1)
  il_6_T2: number analyzed (Participants) | 70 | 66
  il_6_T2 | 0.75 (1.58) | 0.9 (1.97)
  il_6_T3: number analyzed (Participants) | 52 | 56
  il_6_T3 | 0.68 (1.62) | 1.48 (4.11)
  tnfa_T1 | 10.85 (15.36) | 14.27 (23.07)
  tnfa_T2: number analyzed (Participants) | 71 | 65
  tnfa_T2 | 8.007 (4.8) | 9.64 (11.98)
  tnfa_T3: number analyzed (Participants) | 52 | 55
  tnfa_T3 | 7.56 (10.68) | 10.04 (14.49)
  il_10_T1 | 0.43 (1.3) | 0.65 (2.04)
  il_10_T2: number analyzed (Participants) | 71 | 67
  il_10_T2 | 0.19 (0.43) | 0.53 (1.44)
  il_10_T3: number analyzed (Participants) | 54 | 56
  il_10_T3 | 0.34 (0.99) | 0.718 (2.36)
  tgf_b1_T1: number analyzed (Participants) | 115 | 105
  tgf_b1_T1 | 51085 (32095) | 51016 (31641)
  tgf_b1_T2: number analyzed (Participants) | 69 | 64
  tgf_b1_T2 | 48885 (22571) | 47819 (25255)
  tgf_b1_T3: number analyzed (Participants) | 52 | 50
  tgf_b1_T3 | 51447 (34759) | 48178 (23994)

8. Secondary Outcome: Heart Rate Variability
Description: 20 minutes of resting ECG data will be recorded. The participants will be given instructions not to drink coffee or smoke for 3 hours before the lab visit as well as to sit quietly without talking or moving during the ECG recording. These are physiological data without a specific range, however in our study, for example, at T1 in the art therapy group the measurements ranged from 7.56 to 113.28 miliseconds.
Time Frame: Changes will be measured from baseline (T1), after the intervention (8-10 weeks after baseline, T2) and 8 weeks after the intervention ends (T3)
Population: Each row represents the actual number of participants we were able to collect EKG and obtain a good signal, and data was not discarded because of too much noise, or reporting drinking coffee before the measurement,
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Art Therapy | Mandala Group
Number analyzed (Participants) | 115 | 113
miliseconds
  T1 | 32.63 (21.8) | 37.82 (38.8)
  T2: number analyzed (Participants) | 75 | 69
  T2 | 33.13 (20.21) | 31.89 (20.7)
  T3: number analyzed (Participants) | 54 | 59
  T3 | 35.22226363 (40.4) | 33.58334362 (25.6)

ADVERSE EVENTS:
Time Frame: Participants were followed for an average of 20 weeks. Baseline data was collected following signing informed consent, and two weeks before the intervention began (which was 8 weeks long), and until T3, which occurred 8 weeks after the 8-week intervention ended. Having said that, because of the COVID-10 pandemic, and a war, there were several cases in which the intervention started several weeks late due to lockdowns. Thus, some participants were followed for up to 30 weeks.
Description: Team members received categorization of adverse event descriptions and were requested to document them in Redcap.
Arm/Group | Art Therapy | Mandala Group
All-Cause Mortality (participants affected / at risk) | 1/146 | 1/143
Serious Adverse Events (participants affected / at risk) | 8/146 | 6/143
Other Adverse Events (participants affected / at risk) | 16/146 | 15/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Art Therapy (N=146) | Mandala Group (N=143)
disease progression AE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) — disease progression AE
prolonged hospitalization AE (General disorders) | 2 (2) | 1 (1) — The participant is hospitalized due to a health condition
surgery adverse event reporting (Surgical and medical procedures) | 4 (4) | 4 (4) — Entered into an implant removal surgery with infection
Car accident (General disorders) | 1 (1) | 0 (0) — Pain from car accident
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Art Therapy (N=146) | Mandala Group (N=143)
COVID-19 (General disorders) | 3 (3) | 3 (3) — Participant diagnosed with covid and could not continue participation
Side effect from medication or vaccine- not study related (General disorders) | 2 (2) | 0 (0)
In mourning (Social circumstances) | 1 (1) | 1 (1) — Participant relative or close friend died, so did not attend
Stress from family illness (Social circumstances) | 2 (2) | 0 (0)
War (Social circumstances) | 6 (6) | 11 (11) — Participants not attending/ stress from war situation
Injury (General disorders) | 1 (1) | 0 (0) — Participant broke leg
Medication (General disorders) | 1 (1) | 0 (0) — Participant did not provide ECG because of a medication she is taking for pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form: REPAT study protocol (2018-10-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03377816/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03377816/SAP_001.pdf